CLINICAL TRIAL: NCT06951113
Title: Prevalence of Stress Related Mental Health Disorders in Junior Anesthetists and Intensivists in University Hospitals in Cairo
Brief Title: Prevalence of Mental Health Disorders in Junior Anesthetists and Intensivists
Acronym: mental
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FAMSU MS 87/25
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mental health disorders are rapidly growing nowadays and it is well known that people who are subjected to a long term stress are among the highly vulnerable group. Of those, doctors come first specially those working in anesthesia and ICU field owing to the nature of their work where heavy work load, exposure to occupational hazards and competitive environment predominate. More care is needed to identify the magnitude of the ongoing problem and to stand on its determinants to be able to prevent or treat the negative impact on their health and patients as well.

DETAILED DESCRIPTION:
The mental health of physicians is a concern that is gaining popularity and international attention nowadays. Physicians are not immune to mental disorders and even we can say that they are more vulnerable. Mental disorders increases as stress increases, and working as a physician carries stressors like other highly skilled occupations and that unique to the medical field

Work demands are always high and the work environment is relatively poor with insufficient support. They work for long hours with little appreciation and more blaming. Many of them also share the feeling of mental illness stigma that keep them away from seeking help

Usually physicians face most of the stress in their first years of experience that require more learning and working time accompanied by more financial burden with more incidence of mental illness in those working in the frontline as anesthetists and intensivists. Common mental disorders that frequently affect junior anesthetists and intensivists include burn out, anxiety and depression .

Caring for the mental health of physicians goes beyond caring for a colleague, it is a requisite for a powerful functioning health system. Suffering from mental disorders may lead to more sick absences, less productivity, substance abuse and even suicidal thoughts. Patients are at risk of negligence and more medication errors. This requires structured approach to clarify the misinformation regarding physician well-being, and which individual or intervention that should be prioritized.

This is not an easy task as the problem is complex and needs systematic approach to know the magnitude of the problem in reality and study its determinants and put applicable solutions.

ELIGIBILITY:
Inclusion Criteria:

* working as anesthetist or intensivist
* working experience less than or equal 5 years

Exclusion Criteria:

* personality disorders
* psychiatric diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anesthetists and intensivists with working experience ≤5 years working in university hospitals in Cairo between the period from January 2025 to June 2025
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
o Prevalence of mental health disorders ( burnout, anxiety and depression ) | through study completion, an average of 3 months
  o Prevalence of mental health disorders ( burnout, anxiety and depression ) among junior anesthetists and Intensivists working in university hospitals in Cairo.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Elsharnouby, M. D., Study Director — Faculty of medicine, Ain Shams university
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided